CLINICAL TRIAL: NCT04354389
Title: DAS181 for COVID-19: A Phase II Multicenter, Randomized, Placebo-Controlled, Double-Blind Study
Brief Title: DAS181 for STOP COVID-19
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: No COVID-19 in EU countries - Sponsor withdraw in regulatory stage
Sponsor: Ansun Biopharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: DAS181-2-08; 2020-003192-17 (EudraCT Number)
Record Dates: First submitted 2020-04-15; First posted 2020-04-21 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: COVID-19
Keywords: COVID-19; Lower Respiratory Tract Disease; DAS181; SARS-CoV-2; Coronavirus; Hypoxemia; Ansun
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Hypoxia | interventions — oplunofusp

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- DAS181 b.i.d.+ standard local care for COVID-19 (Experimental): 4.5 mg DAS181 b.i.d nebulized inhalation for 10 consecutive days + standard local care for COVID-19
  Interventions: Drug: DAS181
- Placebo+ standard local care for COVID-19 (Placebo Comparator): nebulized inhalation for 10 consecutive days + standard local care for COVID-19
  Interventions: Drug: Placebo
- DAS181 q.d.+ standard local care for COVID-19 (Experimental): 4.5 mg placebo q.d. nebulized inhalation for 10 consecutive days + standard local care for COVID-19
  Interventions: Drug: DAS181

INTERVENTIONS:
Drug: DAS181 — 4.5 mg b.i.d
  Arms: DAS181 q.d.+ standard local care for COVID-19
Drug: Placebo — q.d. or b.i.d.
  Arms: Placebo+ standard local care for COVID-19
Drug: DAS181 — 4.5 mg q.d.
  Arms: DAS181 b.i.d.+ standard local care for COVID-19

SUMMARY:
It is a multicenter, randomized, placebo-controlled, double-blind study. The study population is defined as subjects diagnosed with lower respiratory tract COVID-19 who require supplemental oxygen ≥2 LPM at the time of randomization.

DETAILED DESCRIPTION:
The first stage is randomized, double-blind study to confirm the optimal dose of the study. Twenty-two (n=22) subjects with COVID-19 and clinically significant impairment of respiratory function will be enrolled to evaluate the two dosing regimens (4.5mg-q.d or 4.5mg-b.i.d) of DAS181. At the end of Stage 1, the Sponsor will evaluate the dose regimen based on the safety and efficacy assessments of the data. An optimal dose will be selected to proceed to Stage 2.

The second stage is a randomized, placebo-controlled and double-blind study to expand enrollment with an additional eighty-two (n=82) subjects to provide adequate power to potentially demonstrate statistically significant therapeutic efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Be ≥18 years of age
2. Provide adequate medical history to permit accurate stratification by health status
3. Prior to SARS CoV 2 infection, has no chronic or recurring requirement for supplemental oxygen
4. Have lower respiratory tract infection (LRTI) confirmed by imaging
5. Has laboratory-confirmation of the presence of SARS-CoV-2 in the respiratory tract
6. At the time of randomization, requires supplemental oxygen ≥2 LPM for treatment of hypoxia or pulmonary stress as evidenced by at least one of the following:

   1. Respiratory rate ≥ 30 breaths/min
   2. SpO2 ≤93% at rest
   3. PaO2/FiO2≤300 mmHg
   4. Showing the progression of lung lesions within 24 to 48h by >50%
7. If female, subject must meet one of the following conditions:

   1. Not be of childbearing potential or
   2. Be of childbearing potential and have a negative urine/serum pregnancy test and agrees to practice an acceptable method of contraception
8. Non-vasectomized males are required to practice effective birth control methods
9. Capable of understanding and complying with procedures as outlined in the protocol
10. Provides signed informed consent prior to the initiation of any screening or study-specific procedures

Exclusion Criteria:

1. At the time of randomization, classified as critical (life-threatening) disease
2. Subjects currently receiving any other investigational drug, as part of a clinical trial or under emergency approval for SARS-CoV-2
3. Subjects who are known asthmatic patients or HIV-positive
4. Subjects who are currently receiving inhaled biologics or anti-viral agents
5. Subjects with severe sepsis due to either their SARS-CoV-2 infection or a concurrent viral, bacterial, or fungal infection with vital organ failure or required vasopressors to maintain blood pressure
6. Subjects with Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), or Alkaline Phosphatase (ALP) ≥3x ULN and Total Bilirubin (TBILI) ≥2xULN
7. Female subjects breastfeeding or planning to breastfeed at any time through 30 days after the last dose of study drug.
8. Psychiatric or cognitive illness or recreational drug/alcohol use that, in the opinion of the principal investigator, would affect subject safety and/or compliance.
9. Subjects with known hypersensitivity to DAS181 and/or any of its components.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07-25 (Estimated); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Percent of subjects return to room air (RTRA) | Day 14

SECONDARY OUTCOMES:
Percent of subjects who have recovered | Day 5, 10, 14, 21, 28
  Percent of subjects who reach level 1 of COVID-19 Clinical Classification (discharged or return to normal activity)
Improved COVID-19 Clinical Classification | Day 28
  time to Improved COVID-19 Clinical Classification 1 to 6 (where higher score means worse outcome)
Return To Room Air (RTRA) | Day 10, 21, 28
  Percent of subjects RTRA
Percent of subjects who achieve clinical stability | Day 28
SARS-CoV-2 RNA undetectable | Day 28
  Time to
Clinical Deterioration | Day 28
  Time to
Percent of subjects discharged | Day 14, 21, 28
  Percent of subjects discharge
Death (all cause) | Day 28
  Time to

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Ho, MD, PhD, Study Director — Ansun Biopharma, Inc.
Locations (2):
- Italy (2):
  - Fondazione IRCCS Ca' Granda - Ospedale Maggiore Policlinico, Milan
  - A.O.U Policlinico Di Modena, Modena

IPD SHARING:
Plan to Share IPD: No